CLINICAL TRIAL: NCT02407587
Title: Cortical Activity in Subjects With Unilateral Cochlear Implants and Preserved Ipsilateral Residual Hearing and the Evolution of Temporal Cortex Changes in New Recipients of Cochlear Implants.
Brief Title: Neuroplastic Changes Seen in Cochlear Implants With Preserved Hearing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unresolved issues with a collaborator.
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: R01997
Record Dates: First submitted 2014-09-18; First posted 2015-04-03 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Cochlear Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- unilateral cochlear implants (Experimental): Study Group
  PET scans for the mature patients with unilateral cochlear implants and preserved hearing
  4 states and each state will be repeated 3 times Cochlear implant only Residual hearing only Combination of implant and residual hearing No auditory stimulation
  Interventions: Device: cochlear implants
- Healthy volunteers (No Intervention): 4 states and each state will be repeated 3 times Auditory stimulation Left ear only Auditory stimulation right ear only Binaural auditory stimulation Silence

INTERVENTIONS:
Device: cochlear implants — PET scans for the mature patients with unilateral cochlear implants and preserved hearing
  4 states and each state will be repeated 3 times Cochlear implant only Residual hearing only Combination of implant and residual hearing No auditory stimulation
  Arms: unilateral cochlear implants

SUMMARY:
Investigators hope to study patients with 1 cochlear implant and who have had hearing preservation surgery and compare the changes in the brain of these patients with normal hearing patients by doing a scan of the brain when listening to speech. The information investigators collect may help investigators to understand how the brain learns to hear with a cochlear implant and whether it uses the same areas in the brain to listen as in normal hearing patients as well as predict which patients will do well with a cochlear implant as a very specialised operation is needed to insert the cochlear implant in to the ear and is done by very few surgeons in the country. After the operation, patients need several months of teaching to help them learn how to hear through the implant. Having a cochlear implant requires a lot of cooperation and time from the patient and if investigators could understand how the brain learns to hear with a cochlear implant and predict which patients do well and why then we may be able to avoid unnecessary procedures.

DETAILED DESCRIPTION:
Cochlear implants are an established treatment for individuals with hearing loss where conventional hearing aids fail to provide appropriate hearing amplification and result in poor speech and language perception.

Although a large proportion of patients with cochlear implants are expected to do well with an implant, there is still uncertainty why some individuals do poorly.

Furthermore investigators have limited knowledge about how the brain interacts with a cochlear implant to process speech. Evidence suggests that the underlying central mechanisms responsible for processing speech using an implant are related to neuroplasticity. That is to say that the brain establishes new cortical networks between the vital auditory centres and the cochlear implant thus enabling processing of speech.

Investigators have recently completed a study comparing the cortical changes that occur in subjects with bilateral cochlear implants to normal hearing controls. In this study both groups of patients were subjected to binaural simultaneous auditory stimuli. Analysis suggests that subjects with bilateral cochlear implants and postlingual hearing loss seem to recruit similar areas of the temporal lobes to process speech as their normal hearing counterparts.

The implant recipients activations were larger and more diffuse but did not differ greatly from those described previously in normal hearing. This study provides a good comparison of hearing using bilateral cochlear implants to that of normal unaided hearing. This study provides a more realistic comparison of cortical activations due to hearing in cochlear implantees and normal hearing subjects. This is in contrast to other studies involving monaural stimulation of a unilateral cochlear implant to monaural stimulation of normal hearing subject with the contralateral normal hearing ear blocked off. Investigators are only aware of one additional study where subjects with bilateral cochlear implants have been compared to normal hearing controls.

In addition investigators did not observe any recruitment of the visual cortices in our bilaterally implanted subjects. This finding was also present in Strelnikov's study. However previous work has suggested subjects with cochlear implants rely on visual clues to process speech as a result of the degraded signal provided by the implant. It is possible that because the subjects in this study and Strelnikov's study were experienced implant users and benefited from binaural auditory stimulation, they were not dependant on audio-visual integration to process speech.

There has been an increasing trend towards hearing preservation surgery for patients undergoing cochlear implantation. Literature supports improved speech and pitch perception in quiet and noise for subjects who combine the use of their implant with any residual preserved natural hearing compared with using the implant alone. Once again the the underlying mechanisms for this are unknown. It would be of scientific interest to investigate the interaction between natural residual hearing and hearing via a cochlear implant. It is likely that this cohort of subjects process speech similarly to those with normal hearing.

Finally, studies have monitored the speech progression of implantees from before surgery to several years post implant switch on. It has been suggested that the predominant improvement in speech perception occurs in the first year of implant use. This would suggest that the neuronal networks responsible for speech processing are established very early on however, investigators are not aware of any studies which have attempted to track the evolution of the temporal cortices in new recipients of cochlear implants.

ELIGIBILITY:
Inclusion Criteria:

* Mature users of unilateral cochlear implants who have natural preserved hearing in the implanted ear
* Healthy volunteers with normal hearing
* Right handed

Exclusion Criteria:

* Individuals with neurological or psychiatric illness
* Patients involved in additional drug trials
* Pregnant or breast feeding women
* Children
* Left-handed subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05 (Estimated); Primary Completion 2015-10 (Estimated); Study Completion 2017-02-27 (Actual)

PRIMARY OUTCOMES:
Increase our understanding of why outcomes following a cochlear implant are heterogenous. This information may be used to provide targeted rehabilitation for candidates performing poorly with their implants and minimise rejection of the implant. | 1 year
  We anticipate that the recruitment of patients, data collection and analysis would take a maximum of 4 months
  Study Group
  PET scans for the mature patients with unilateral cochlear implants and preserved hearing
  4 states and each state will be repeated 3 times Cochlear implant only Residual hearing only Combination of implant and residual hearing No auditory stimulation
  Control Group
  4 states and each state will be repeated 3 times Auditory stimulation Left ear only Auditory stimulation right ear only Binaural auditory stimulation Silence

SECONDARY OUTCOMES:
Combine the data from both of our studies and future studies in order to conduct meta-analysis to investigate further how language is processed in patients with cochlear implants. | 1 year
Determine if functional neuroimaging modalities have a future role in the selection process for potential cochlear implant candidates and in predicting outcome for each individual. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rohini Aggrawal, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Central Manchester University Hospitals NHS Foundation Trust, Manchester, Manchester (Manchester Borough), United Kingdom